CLINICAL TRIAL: NCT00062647
Title: A Phase 2, Randomized, Double-Blind, Parallel-Group, Multinational Trial of Intravenous Televancin (TD-6424) for Treatment of Uncomplicated Staphylococcus Aureus Bacteremia
Brief Title: Telavancin for Treatment of Uncomplicated Staphylococcus Aureus Bacteremia
Acronym: ASSURE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Steven L. Barriere, Pharm.D., Vice President, Clinical and Medical Affairs, Theravance, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: I6424-203a
Record Dates: First submitted 2003-06-09; First posted 2003-06-12 (Estimated); Results first posted 2011-03-22 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Gram-Positive Bacterial Infections
MeSH Terms: conditions — Gram-Positive Bacterial Infections | interventions — telavancin; Vancomycin; Nafcillin; Oxacillin; Cloxacillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telavancin (Experimental)
  Interventions: Drug: Telavancin
- Vancomycin, nafcillin, oxacillin, or cloxacillin (Active Comparator): Vancomycin 1 Gram/12 hours or nafcillin, oxacillin, or cloxacillin 2 Gram/6 hours (IV) intravenously
  Interventions: Drug: Vancomycin, nafcillin, oxacillin, or cloxacillin

INTERVENTIONS:
Drug: Telavancin — Telavancin 10mg/kg/day IV every 24 hrs for up to 14 days
  Other Names: TD-6424; VIBATIV
  Arms: Telavancin
Drug: Vancomycin, nafcillin, oxacillin, or cloxacillin — Vancomycin 1 Gram every 12 hr IV (intravenously) OR nafcillin, oxacillin, or cloxacillin 2 Grams every 6 hr IV (intravenously) for up to 14 days.
  Arms: Vancomycin, nafcillin, oxacillin, or cloxacillin

SUMMARY:
The purpose of this study is to determine whether telavancin (TD-6424, ARBELIC) can be safety administered to patients with bloodstream infections and whether telavancin is effective in treating these infections.

ELIGIBILITY:
Inclusion Criteria

- Documented S. aureus bacteremia

Exclusion Criteria

- Patients who had received or would have received more than 72 hours of potentially effective systemic antistaphylococcal therapy within 7 days prior to randomization. The following agents were considered potentially effective antistaphylococcal therapy: antistaphylococcal penicillins (including nafcillin, oxacillin, or cloxacillin), cephalosporins, fluoroquinolones, glycopeptides (including vancomycin and teicoplanin) and linezolid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-08; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G. Ralph Corey, MD, Principal Investigator — Duke University
Locations (1):
- Wellstar Infectious Disease, Marietta, Georgia, United States

REFERENCES:
- [Derived] Stryjewski ME, Lentnek A, O'Riordan W, Pullman J, Tambyah PA, Miro JM, Fowler VG Jr, Barriere SL, Kitt MM, Corey GR. A randomized Phase 2 trial of telavancin versus standard therapy in patients with uncomplicated Staphylococcus aureus bacteremia: the ASSURE study. BMC Infect Dis. 2014 May 23;14:289. doi: 10.1186/1471-2334-14-289. PMID 24884578

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period: 14 Aug 2003 to 02 Aug 2006
Groups:
- Telavancin: Patients with uncomplicated Staphylococcus aureus bacteremia were randomized to receive telavancin 10 mg/kg/day IV (intravenously) every 12 hrs for up to 14 days. Excludes 1 patient who never started therapy.
- Standard Therapy: Patients with uncomplicated Staphylococcus aureus bacteremia were randomized to receive vancomycin 1 Gram IV (intravenously) every 12 hrs OR nafcillin, oxacillin, or cloxacillin 2 Gram IV (intravenously) every 6 hrs for up to 14 days. Excludes one patient who never started therapy.
Period: Overall Study
Arm/Group | Telavancin | Standard Therapy
Started | 30 | 30
Completed | 14 | 17
Not Completed | 16 | 13
Not completed — Death | 2 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Failed continuation criteria | 4 | 2
Not completed — Other | 4 | 4
Not completed — Never received study treatment | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telavancin | Standard Therapy | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (19) | 60 (17.9) | 60 (17.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 18 | 15 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 22 | 22 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 3 | 12
  White | 17 | 21 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 3 | 2 | 5
  Singapore | 1 | 3 | 4
  Spain | 2 | 3 | 5
  United States | 22 | 21 | 43
  Hong Kong | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response (Cure, Failure, or Indeterminate) as Determined by the Investigator Based the Presence or Absence of Clinical Signs and Symptoms Associated With Bacteremia, Metastatic Complications, or Positive Culture at the Test of Cure Evaluation
Description: Outcomes in this exploratory study were compared for noninferiority though no specific margin was justified. The 95% CI for the difference was -35.5 to 31.9; further statistical evaluation is not warranted owing to the small sample size.
Time Frame: 12 weeks after start of treatment
Population: The primary efficacy analysis was of the CE Population, defined as those patients meeting meeting inclusion/exclusion criteria, meeting continuation criteria, receiving assigned study drug for at least 14 days and available for assessment of response.
Measure: Number; unit: participants
Arm/Group | Telavancin | Standard Therapy
Number analyzed (Participants) | 8 | 9
participants
  Cured | 7 | 8
  Failure | 1 | 1
Statistical Analysis 1: Comparison: Telavancin vs Standard Therapy; Test type: Non-Inferiority or Equivalence — No margin was justified owing to the exploratory nature of the investigation; the difference in the 2 eradication rate; Statistical testing was limited to interval estimation (95% CI) of the difference in the 2 eradication rates using the method of Agresti and Caffo; Risk Difference (RD) = 1, 95% CI [-35.5 to 31.9]

ADVERSE EVENTS:
Time Frame: From receipt of first dose through last follow-up assessment (up to Day 98).
Arm/Group | Telavancin | Standard Therapy
Serious Adverse Events (participants affected / at risk) | 11/29 | 6/29
Other Adverse Events (participants affected / at risk) | 26/29 | 21/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telavancin (N=29) | Standard Therapy (N=29)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse Drug Reaction (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Multi-organ Failure (General disorders) | 1 (1) | 1 (1)
Neuroleptic Malignant Syndrome (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis bacterial (Cardiac disorders) | 1 (1) | 0 (0)
Lobar Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure Chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telavancin (N=29) | Standard Therapy (N=29)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Catheter site erythema (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 2 (2)
Catheter site infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary Tract Infection Fungal (Infections and infestations) | 2 (2) | 0 (0)
Blood Urea increased (Investigations) | 2 (2) | 0 (0)
Eosinophil Count increased (Investigations) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Agitation (Psychiatric disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Deep Vein Thrombosis (Vascular disorders) | 3 (3) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less